CLINICAL TRIAL: NCT01289899
Title: BR-A-657, A Phase 1, Double-blind, Placebo-controlled, Ascending Multiple Oral Dose Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study in Healthy Male Subjects
Brief Title: Fimasartan (BR-A-657) Multiple Oral Dose in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Covance (Industry)
Responsible Party: Paik, Assistant manager, Boryung Pharm. Co., Ltd
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2290/9
Record Dates: First submitted 2010-12-14; First posted 2011-02-04 (Estimated); Last update posted 2011-02-04 (Estimated); Status verified 2011-02

CONDITIONS: Essential Hypertension
Keywords: BR-A-657; Fimasartan; multiple-dose; pharmacokinetic; pharmacodynamic; safety
MeSH Terms: conditions — Essential Hypertension | interventions — fimasartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): BR-A-657 120mg or placebo
  Interventions: Drug: BR-A-657
- Arm B (Experimental): BR-A-657 360mg or placebo
  Interventions: Drug: BR-A-657

INTERVENTIONS:
Drug: BR-A-657 — 120, 360mg or placebo 7days
  Other Names: Fimasartan

SUMMARY:
The objective of this study is to determine the safety and tolerability and to determine the Pharmacokinetic and Pharmacodynamic(PK/PD) of ascending multiple oral dose of BR-A-657 in healthy male subjects.

DETAILED DESCRIPTION:
BR-A-657 120, 360, or placebo were administered once daily for 7days to 16 healthy male subjects.

Pharmacokinetic and Pharmacodynamic(PK/PD) parameters were monitored at pre-specified times from each subjects.

PK parameters: Area Under the Curve(AUC), Cmax, half-life, etc. PD parameters: Aldosterone, Plasma renin activity, Angiotensin I, Angiotensin II Adverse events are reported.

ELIGIBILITY:
Inclusion Criteria:

* male of 18-55 years old
* BMI 19-29kg/m2
* subjects in good health
* subjects with written informed consent

Exclusion Criteria:

* subjects with multiple drug allergy or allergy to ARB
* subjects with medication that affect drug absorption or elimination within 30days.
* subjects with orthostatic hypotension of >20mmHg decrease of sbp
* subjects with history of neurologic, liver, renal, GI, CV, psychological or other major disorder

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2004-01; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
No of subjects with Adverse events(AE) from each observations | up to 5~7days post final(7th) dose
  1. AE reporting: Day 1: Predose, 3 & 12h, Days 2~7: Predose, Days 8,9: Once daily, 5~7days post final dose
  2. Vital signs: Day 1: Predose, 0.5,1,2,4,8,12,24h,Days 3~6: Predose Day 7: Predose, 0.5,1,2,4,8,12,24,48h, 5~7days post final dose
  3. ECG: Days 1 & 7: Predose, 2, 4, 8 & 24h, Day 4: Predose, 5~7days post final dose
  4. Laboratory examination: Days 1 & 4: Predose, Day 7: Predose & 24h, 5~7days post final dose
  5. Physical examination: predose, 5~7days post final dose
  6. Body weight: predose, Days 4 & 8

SECONDARY OUTCOMES:
Area under the plasma concentration time curve (AUC) | predose,0.5,1,1.5,2,3,4,6,8,12,16,24,(48)h on day 1 and day 7
Maximum observed plasma concentration (Cmax). | predose,0.5,1,1.5,2,3,4,6,8,12,16,24,(48)h on day 1 and day 7
parent plasma terminal elimination half life (t½) | predose,0.5,1,1.5,2,3,4,6,8,12,16,24,(48)h on day 1 and day 7
Apparent total plasma clearance (CL/F) | predose,0.5,1,1.5,2,3,4,6,8,12,16,24,(48)h on day 1 and day 7
Accumulation ratio (RA) | predose,0.5,1,1.5,2,3,4,6,8,12,16,24,(48)h on day 1 and day 7
  RA1=Accumulation ratio based on AUCinf
  RA2=Accumulation ratio based on Cmax

CONTACTS AND LOCATIONS:
Overall Officials: E Engmann, MB ChB, Principal Investigator — Covance Clinical Research Unit